CLINICAL TRIAL: NCT00998660
Title: RECHARGE Sub-Study to the Implantable Systems Performance Registry (ISPR)
Acronym: RECHARGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1649
Record Dates: First submitted 2009-10-12; First posted 2009-10-20 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease; Essential Tremor; Dystonia
Keywords: Parkinson's disease; Essential Tremor; Dystonia (where indication is approved); Deep brain stimulation; Activa RC
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients receiving an Activa RC implant (Experimental)
  Interventions: Device: Activa RC

INTERVENTIONS:
Device: Activa RC — Patients receiving Activa RC as their first implantable neurostimulator or as a replacement implantable neurostimulator for deep brain stimulation

SUMMARY:
The purpose of this study is to assess the recharge feature of the Activa RC System in patients who are receiving Deep Brain Stimulation (DBS) for Parkinson's Disease (PD), Essential Tremor (ET), or dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Patient is enrolled in the Implantable Systems Performance Registry (ISPR) and will receive one Activa RC as their first implantable neurostimulator or as a replacement implantable neurostimulator for DBS.
* Patient must meet the indications in the Activa RC labeling.
* Patient (or patient's legally authorized representative) signs and dates the appropriate RECHARGE Informed Consent Form and/or Informed Assent Form and Authorization to Use and Disclose Health Information (HIPAA, US only).
* Patient has a diagnosis of Parkinson's Disease, Essential Tremor, or dystonia that meets the approved indication for Activa RC in the applicable geography.
* Patient with dystonia is 7 years of age or older (EU only).
* Patient with either PD or ET is 18 years of age or older.
* Patient (or caregiver) is able to use the patient programmer and correctly interpret the icons.
* Patient (or caregiver) is able and willing to regularly monitor the status of the rechargeable battery and respond appropriately.
* Patient (or caregiver) is able to locate the INS, position the recharge antenna for sufficient coupling, put on the recharge holster/belt, and monitor progress during the recharge session.
* Patient (or caregiver) is able to perform recharging activities for sufficient duration and frequency to maintain therapy and to perform recharging activities on an ongoing basis.
* Patient is willing and able to comply with protocol requirements.

Exclusion Criteria:

* Patient has a contraindication identified in the Activa RC labeling.
* Patient who is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound the results of the RECHARGE study.
* Patient has or will be implanted with a non-Medtronic Deep Brain Stimulation system component.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ISPR Team, Study Chair — Medtronic
Locations (11):
- United States (5):
  - Washington D.C., District of Columbia
  - Cincinnati, Ohio
  - Nashville, Tennessee
  - Houston, Texas
  - Tyler, Texas
- Vienna, Austria
- Montpellier, France
- Germany (2):
  - Cologne
  - Hanover
- Barcelona, Spain
- Oxford, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Receiving an Activa RC Implant
Started | 100
Implanted | 93
Month 3 Visit | 87
Completed | 87 (87 subjects reached the final study visit at Month 6.)
Not Completed | 13

BASELINE CHARACTERISTICS:
Groups:
- Dystonia Patients Implanted With the Activa RC: Patients who were implanted with the Activa RC neurostimulator to treat dystonia.
- Essential Tremor Patients Implanted With the Activa RC: Patients who were implanted with the Activa RC neurostimulator to treat Essential Tremor.
- Parkinsons Disease Patients Implanted With the Activa RC: Patients who were implanted with the Activa RC neurostimulator to treat Parkinson's Disease.
- Total: Total of all reporting groups
Arm/Group | Dystonia Patients Implanted With the Activa RC | Essential Tremor Patients Implanted With the Activa RC | Parkinsons Disease Patients Implanted With the Activa RC | Total
Number analyzed (Participants) | 28 | 11 | 54 | 93
Age, Continuous [Mean (Full Range); unit: years] | 40.4 [11 to 82] | 64.5 [39 to 79] | 59.6 [39 to 79] | 54.4 [11 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 11 | 31
  Male | 15 | 4 | 43 | 62
Region of Enrollment [Number; unit: participants]
  United States | 0 | 10 | 35 | 45
  France | 15 | 0 | 0 | 15
  Spain | 1 | 0 | 1 | 2
  Austria | 5 | 0 | 4 | 9
  Germany | 6 | 1 | 10 | 17
  United Kingdom | 1 | 0 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Identify the Rate of User-related Battery Depletion Adverse Events Per Subject-month Requiring Intervention by a Health Care Professional (HCP) and/or the HCP's Designee, Within the First 3 Months of the Activa RC System Being Turned ON.
Description: Subject-months of follow-up were defined as the time from device activation to the earlier of a subject's 3-month visit or until the subject exited from the study. Any user-related battery depletion adverse events requiring intervention by a health care professional (HCP) and/or the HCP's designee were collected. The event rate per 100 subject-months of follow-up is defined as the number of user-related battery depletion events divided by the total subject follow-up months through the 3-month visit, all multiplied by 100.
Time Frame: 3 months
Population: The 93 implanted subjects accumulated 283.6 subject-months of follow-up through the 3-month visit. There were no reported user-related battery depletion adverse events that required an intervention by a health care professional and/or HCP designee.
Measure: Number (95% Confidence Interval); unit: Event rate per 100 subject-months
Groups:
- Patients Implanted With the Activa RC: All enrolled patients implanted with the Activa RC neurostimulator.
Arm/Group | Patients Implanted With the Activa RC
Number analyzed (Participants) | 93
Event rate per 100 subject-months | 0.00 [0.00 to 1.30]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Activa RC implant through discontinuation (maximum of 6 months).
Description: The occurrence of adverse events was assessed by the investigator at each study visit. All adverse events, regardless of relatedness to the device and/or therapy, were collected. Within the 93 implanted subjects, there was 560.4 months of study follow-up from Activa RC implant to study discontinuation.
Arm/Group | Patients Implanted With the Activa RC
Serious Adverse Events (participants affected / at risk) | 9/93
Other Adverse Events (participants affected / at risk) | 0/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Implanted With the Activa RC (N=93)
Dyskinesia (Nervous system disorders) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1)
Implant site inflammation (General disorders) | 1 (1)
Implant site pain (General disorders) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Potential limitations of the study include the limited sample size to fully characterize recharge use by indication. In addition, inferences to a broader population should also be limited given the relatively short duration of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will review results communications prior to public release to determine whether Confidential Information is disclosed and will not censor or in any way interfere with presentation or conclusions beyond the extent necessary to protect Confidential Information. PIs are required to provide results communications for review at least 60 days prior to submission or presentation. When requested by Sponsor, PI will delay publication up to an additional 90 days.